CLINICAL TRIAL: NCT05499117
Title: Efficacy and Safety of Light Therapy in the Treatment of Non-seasonal Depressive
Brief Title: Efficacy and Safety of Light Therapy in the Treatment of Non-seasonal Depressive Disorder in Chinese Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-HY-006
Record Dates: First submitted 2022-08-11; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antidepressant and light treatment group (Active Comparator)
  Interventions: Device: Light terapy
- Antidepressants and pseudo-light therapy (Placebo Comparator)
  Interventions: Device: pseudo-light therapy

INTERVENTIONS:
Device: Light terapy — Carex Day-Light Classic, Light intensity is white Light, 10000UX, and color temperature is 4000K
  Other Names: fluoxetine
  Arms: Antidepressant and light treatment group
Device: pseudo-light therapy — The pseudo-light stimulation group was red light with intensity less than 100lux
  Other Names: fluoxetine
  Arms: Antidepressants and pseudo-light therapy

SUMMARY:
Depression is a kind of mental illness with high incidence, high recurrence and high disability. But so far, treatment remission rates for depression remain low. Therefore, it is necessary to develop more new treatments. Light therapy has been shown to be effective in treating depression with seasonal patterns. Although most studies have reported that light therapy is also effective in patients with depression without seasonal patterns, high-quality clinical studies are still rare and the conclusions are still controversial. In particular, it remains unclear whether light therapy is effective in treating depression without seasonal patterns in the Chinese population. In addition, there is a lack of biomarkers that predict the efficacy of light therapy.

In conclusion, this study intends to conduct an ADD-ON randomized controlled study to clarify the efficacy and safety of light therapy as synergistic therapy in patients with depression without seasonal patterns, and to screen peripheral biomarkers related to efficacy using transcriptome sequencing technology. It is expected that this study can confirm the effectiveness and safety of light therapy as synergistic therapy, provide an evidence-based basis for the research and exploration of light therapy in Chinese depression population, and provide more options for the synergistic treatment of antidepressants in Chinese depression population.

ELIGIBILITY:
Inclusion Criteria:

1）Meets DSM-5 criteria for major depressive disorder 2) Age 18-65; 3) HAMD-17 score ≥17; 4) No antidepressants or mood stabilizers were used at least 2 weeks before enrollment; 5) Sign informed consent.

Exclusion Criteria:

1. With seasonal pattern;
2. No previous mental disorders, personality disorders, mental retardation, neurodegenerative diseases, brain trauma, cerebrovascular diseases caused by organic diseases;
3. No previous history of alcohol or substance dependence;
4. Current serious risk of suicide (e.g., previous attempted suicide or recent suicidal behavior); 5）Present with serious, active physical diseases that may interfere with research, including vision problems and photosensitivity disorders; 6）Have received electroconvulsive therapy (ECT or MECT) or transcranial magnetic stimulation (rTMS) in the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
remission of acute phase | 8 weeks
  scored 7 or lower on the Hamilton's Depression Scale with 17 items

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided